CLINICAL TRIAL: NCT03617328
Title: Evaluation of Safety and Durable Immunogenicity of Melanoma Vaccination, With or Without Systemic CDX-1127, in Patients With Stage II-IV Melanoma
Brief Title: Vaccination With 6MHP, With or Without Systemic CDX-1127, in Patients With Stage II-IV Melanoma
Acronym: Mel-65
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor of Surgery; Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20085
Record Dates: First submitted 2018-06-28; First posted 2018-08-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Melanoma
Keywords: peptide; vaccine; adjuvant; 6MHP; polyICLC; varlilumab; CDX-1127; Montanide ISA-51
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51; varlilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: 6MHP/Montanide ISA-51 + polyICLC + CDX-1127 (Experimental): 200 mcg of 6MHP plus 0.9 mg of polyICLC emulsified in Montanide ISA-51 adjuvant will be administered subcutaneously on days 1, 8, 15, and 36. 200 mcg of 6MHP in Montanide ISA-51 adjuvant (without polyICLC) will be administered subcutaneously/intradermally on day 176. CDX-1127 (3mg/kg) will be administered intravenously on days 1, 36, and 78.
  Interventions: Biological: 6MHP; Drug: Montanide ISA-51; Drug: polyICLC; Drug: CDX-1127
- Arm B: 6MHP/Montanide ISA-51 + polyICLC (Experimental): 200 mcg of 6MHP plus 0.9 mg of polyICLC emulsified in Montanide ISA-51 adjuvant will be administered subcutaneously on days 1, 8, 15, and 36. 200 mcg of 6MHP in Montanide ISA-51 adjuvant (without polyICLC) will be administered subcutaneously/intradermally on day 176.
  Interventions: Biological: 6MHP; Drug: Montanide ISA-51; Drug: polyICLC

INTERVENTIONS:
Biological: 6MHP — 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Other Names: 6 melanoma helper peptide vaccine
Drug: Montanide ISA-51 — Montanide ISA-51 (Incomplete Freund's Adjuvant), local adjuvant
Drug: polyICLC — polyICLC, local adjuvant
Drug: CDX-1127 — CDX-1127, anti-CD27 monoclonal antibody
  Other Names: Varlilumab
  Arms: Arm A: 6MHP/Montanide ISA-51 + polyICLC + CDX-1127

SUMMARY:
This study evaluates whether it is safe to administer a peptide vaccine (6MHP) with adjuvants and the CDX-1127 monoclonal antibody, and whether the adjuvants and the CDX-1127 monoclonal antibody boost immune responses to the vaccine. In this study, the adjuvants are Montanide ISA-51 and polyICLC. The investigators will monitor these effects by performing tests in the laboratory on participants' blood and tissue from a vaccine site.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patients with stage IIB, IIC, III, or IV melanoma at original diagnosis or at restaging after recurrence, rendered clinically free of disease by surgery, other therapy, or spontaneous remission within 6 months prior to registration.
2. Patients with small radiologic or clinical findings of an indeterminate nature may be eligible.
3. Patients with high-risk stage IIA melanoma (by DecisionDx Melanoma test, Castle Biosciences, Inc., Friendswood, TX) may be eligible.
4. Participants may have had cutaneous, uveal, mucosal primary melanoma, or an unknown primary melanoma. Diagnosis of melanoma must be confirmed by cytological or histological examination. Staging of cutaneous melanoma will be based on version 8 AJCC staging system.
5. Participants who have had brain metastases will be eligible if all of the following are true:

   * Each brain metastasis must have been completely removed by surgery or each unresected brain metastasis must have been treated with stereotactic radiosurgery.
   * No brain metastasis is > 2 cm in diameter at the time of registration.
   * Any neurologic symptoms attributable to brain metastases have returned to baseline.There is no evidence of new or enlarging brain metastases.
   * The most recent surgical resections or gamma-knife therapy for malignant melanoma must have been completed ≥ 1 week and ≤ 6 months prior to registration.
6. ECOG performance status of 0 or 1.
7. Ability and willingness to give informed consent.
8. Adequate organ function
9. Age 18 years or older at registration.

Main Exclusion Criteria:

1. The following medications or treatments at any time within 4 weeks of registration:

   * Chemotherapy
   * Interferon (e.g. Intron-A®)
   * Radiation therapy (Stereotactic radiotherapy, such as gamma knife, can be used ≥ 1 week and ≤ 6 months prior to registration)
   * Allergy desensitization injections
   * High doses of systemic corticosteroids
   * Growth factors (e.g. Procrit®, Aranesp®, Neulasta®)
   * Interleukins (e.g. Proleukin®)
   * Any investigational medication
   * Targeted therapies specific for mutated BRAF or for MEK
2. Nitrosoureas within 6 weeks of registration.
3. Checkpoint molecule blockade therapy within 12 weeks of registration.
4. Known or suspected allergies to any component of the vaccine.
5. Previous vaccination with 6MHP.
6. Prior treatment with CDX-1127 or other CD27 agonistic antibody.
7. Pregnancy.
8. HIV positivity or evidence of active Hepatitis C virus.
9. Female participants must not be breastfeeding.
10. A medical contraindication or potential problem in complying with the requirements of the protocol in the opinion of the investigator.
11. New York Heart Association classification as having Class III or IV heart disease.
12. Uncontrolled diabetes, defined as having an HgbA1c > 8.5%.
13. Prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded.
14. Participants with known addiction to alcohol or drugs who are actively taking those agents, or participants with recent (within 1 year) or ongoing illicit IV drug use.
15. Participants who have received a live vaccine within 30 days of registration.
16. Body weight < 110 pounds at registration, due to the amount and frequency with which blood will be drawn.
17. Participants with prior autoimmune pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Safety of CDX-1127 administered with a melanoma vaccine | 30 days after receiving the last dose of study drug
  Number of participants with dose-limiting toxicities based on CTCAE v5.0
Immunogenicity-Percent of patients with persistent CD4+ T cell responses to the 6MHP vaccine | Day 127 or Day 176 or both
  Number of participants with CD4+ T cell responses to 6 MHP persisting to day 127 or later.

SECONDARY OUTCOMES:
Immunologic effect of CDX-1127 - Impact on regulatory T cells | Day 22 and Day 85 (Note: Day 85 biopsy not required for participants whose Day 85 visit would be due after IRB approval of Protocol v12-03-2020)
  Number of regulatory T cells per mm2 in the vaccine site microenvironment
Immunologic effect of CDX-1127 - Percent of circulating regulatory T cells | through day 176
  Percent of circulating regulatory T cells among CD4+ T cells
Immunogenicity - Frequency of circulating CD4+ Th1 responses | through day 176
  Number of participants with circulating CD4+ Th1 responses to vaccine antigens
Immunogenicity-Frequency of durable CD4+ Th1 memory responses | Day 8 to Day 85
  Number of participants with durable CD4+ Th1 memory response to vaccine antigens, measured as response at two or more consecutive time points
Immunogenicity-Frequency of CD4+ Th1 memory responses | Day 183
  Number of participants with CD4+ Th1 memory response to vaccine antigens a week after the Day 176 booster vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, Jr., MD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared starting 1 year after publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 1 year after publication
Access Criteria: The PI will review access requests. We may share files or share documents through a shared server.